CLINICAL TRIAL: NCT04989218
Title: An Open-label Window of Opportunity Trial to Evaluate the Activity of Durvalumab (MEDI4736) and Tremelimumab With Platinum-based Chemotherapy (Gemcitabine and Cisplatin) in Intrahepatic Cholangiocarcinoma (ICC)
Brief Title: Durvalumab and Tremelimumab With Platinum-based Chemotherapy in Intrahepatic Cholangiocarcinoma (ICC)
Acronym: ICC
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Slow accrual and study sponsor decision.
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Mehmet Akce, MD, Associate Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300005453; 000538122 (Other Grant/Funding Number: Astra Zeneca)
Record Dates: First submitted 2021-07-09; First posted 2021-08-04 (Actual); Results first posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Cholangiocarcinoma
Keywords: Durvalumab; Tremelimumab; Platinum-based chemotherapy; Gemcitabine; Cisplatin
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Immunotherapy; Cisplatin; Gemcitabine; durvalumab; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Novel combination of chemotherapy and immunotherapy (Experimental): This study has one arm. All enrolled patients will receive a combination of a platinum based chemotherapy regimen (gemcitabine and cisplatin) and a combination of two immune check point inhibitors, anti- CTLA4 (Tremelimumab) and anti PDL-1 (durvalumab).
  Gemcitabine will be administered (gemzar) intravenously, 1000mg/m2 on Day 1 and Day 8 of a 21 day cycle for up to 4 cycles. Cisplatin (Platinol) will be administered intravenously, 25mg//m2 on Day 1 and Day 8 of a 21 day cycle for up to 4 cycles.
  Tremelimumab will be administered intravenously, 300mg flat dose, on Day 1 of cycle 1 only. Durvalumab will be administered intravenously 1500mg on Day 1 of a 21 day cycle for 4 cycles.
  Interventions: Drug: Novel combination of chemotherapy and immunotherapy

INTERVENTIONS:
Drug: Novel combination of chemotherapy and immunotherapy — This is a study of the combination of platinum based chemotherapy (gemcitabine and cisplatin) and doublet immunotherapy (durvalumab and tremelimumab) in the preoperative setting for intrahepatic cholangiocarcinoma with high risk features. Gemcitabine and cisplatin are chemotherapy agents used in the management of locally advanced and metastatic cholangiocarcinoma. Durvalumab is a programmed cell death ligand 1 (PDL1) blocking antibody, that improves the immune response against cancer. Tremelimumab is an antibody that targets cytotoxic T cell lymphocyte-associated protein 4 (CTLA4) on regulatory T cells. It also improves the immune response against cancer cells
  Other Names: Cisplatin (Platinol); Gemcitabine (Gemzar); Durvalumab (Imfimzi); Tremelimumab

SUMMARY:
This pilot trial will be used to assess the activity, safety and feasibility of doublet immunotherapy and platinum-based chemotherapy in resectable intrahepatic cholangiocarcinoma with high risk features. The hypothesis is that the combination of durvalumab/MEDI4736 and tremelimumab (doublet immunotherapy) with platinum-based chemotherapy (gemcitabine and cisplatin) will yield an objective of 52% and improve complete resection rates in intrahepatic cholangiocarcinoma. This will facilitate margin negative resection and ultimately reduce recurrence rates and improve survival. Carrying out this trial in the neoadjuvant setting potentially allows improved overall survival and also provides an opportunity for discovery of biomarkers that may predict response to therapy.

DETAILED DESCRIPTION:
All enrolled participants will receive the study intervention. Patients will receive up to 4 cycles of interventional agents prior to surgical resection. They will undergo imaging scans after the 2nd and 4th cycle (before surgery) of intervention agents. The short interval of scans (6 weeks) allows investigators to identify non responders. These patients may be encouraged to come off study and be treated based on the treating oncologist's choice. Since the investigational agents include 'standard of care' agents, a good argument can be made that these patients would not have benefitted from standard therapy only. Patients with at least stable disease after the 2nd treatment cycle will proceed with study interventions. However, patients with radiologic progression but who remain clinically stable may be allowed to continue treatment if the patient elects to, pending confirmation of progression and after a discussion between the investigator and sponsor-investigator.

ELIGIBILITY:
Inclusion Criteria:

Subject must meet all of the following applicable inclusion criteria to participate in this study:

1. Histologically/cytologically confirmed diagnosed intrahepatic cholangiocarcinoma
2. Measurable disease based on RECIST 1.1 and have 1 or more radiologic features compatible with high risk (for resection and recurrence) but still considered technically resectable per multidisciplinary tumor board (Surgical oncologist, radiologist and medical oncologist minimum) meeting. High risk features would include at least 1 of the following criteria-

   • A large tumor (> 5cm) that would benefit from preoperative tumor shrinkage with systemic therapy
   * T1b-T4 tumor thought to be technically resectable
   * Multifocal tumors/ a tumor with satellite lesions confined to the same lobe, thought to be technically resectable
   * Suspicious or involved lymph nodes (N1) thought to be technically resectable
   * Tumor with any vascular involvement/invasion considered technically resectable
   * No extrahepatic metastases
3. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. Written informed consent and any locally required authorization (e.g., Health Insurance Portability and Accountability Act in the US) obtained from the patient/legal representative prior to performing any protocol-related procedures, including screening evaluations.
4. Adult male or female age >18 years at time of study entry
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
6. Life expectancy of > 6 months
7. Body weight >30 kg
8. Adequate normal organ and marrow function as defined below:

   * Hemoglobin ≥ 10.0 g/dL
   * Absolute neutrophil count (ANC ≥1.5 x 109/L (> 1500 per mm3)
   * Platelet count ≥100 x 109/L (>75,000 per mm3)
   * Serum bilirubin ≤1.5 x institutional upper limit of normal (ULN). This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with the sponsor.
   * AST (SGOT)/ALT (SGPT) ≤2.5 x institutional upper limit of normal Measured creatinine clearance (CL) >60 mL/min or Calculated creatinine clearance CL>60 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance
9. Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrhoeic for 12 months without an alternative medical cause. The following age-specific requirements apply:

   * Women <50 years of age would be considered post-menopausal if they have been amenorrhoeic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
   * Women ≥50 years of age would be considered post-menopausal if they have been amenorrhoeic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
10. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
11. Provide archival tumour tissue sample or newly obtained core or excisional biopsy of a previously unirradiated tumour lesion. Tissue blocks are preferred but unstained cut slides acceptable. In addition, should be open to undergoing a biopsy after at least 2 cycles of therapy. Patients who do not undergo surgical resection after 4 cycles will be advised to undergo another biopsy.

Exclusion Criteria:

1. Has had previous local (surgery, radiation, embolizing procedure) or systemic therapy for borderline resectable intrahepatic cholangiocarcinoma.
2. Participation in another clinical study with an investigational product during the last 3 months.
3. Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study.
4. Has ampullary cancer, extrahepatic cholangiocarcinoma or gall bladder cancer.
5. Patients with distant extrahepatic metastatic disease including distant (non-regional lymph nodes). NOTE: Regional lymph nodes depend on tumor site; for left sided lesions, regional lymph nodes include inferior phrenic, hilar and gastrohepatic lymph nodes. For right sided lesions, regional lymph nodes include hilar periduodenal and peripancreatic lymph nodes.
6. Has any other histologic subtype except adenocarcinoma or mixed histology with adenocarcinoma/hepatocellular carcinoma.
7. Any unresolved toxicity NCI CTCAE Grade > 2 from previous anticancer therapy except for alopecia, vitiligo and the laboratory values defined in the inclusion criteria.
8. Patients with Grade ≥ 2 neuropathy will be evaluated on a case-by-case basis after consultation with the sponsor-investigator.
9. Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab or tremelimumab may be included only after consultation with the sponsor-investigator. Any medical contraindication to the use of platinum-based doublet chemotherapy as judged by the treating physician.
10. . Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of study drugs.
11. History of allogenic organ transplantation.
12. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.]). The following are exceptions to this criterion:

    • Patients with vitiligo or alopecia

    • Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
    * Any chronic skin condition that does not require systemic therapy
    * Patients without active disease in the last 5 years may be included but only after consultation with the study physician
    * Patients with celiac disease controlled by diet alone
13. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhoea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent.
14. History of active primary immunodeficiency.
15. History of another primary malignancy except for

    • Malignancy treated with curative intent and with no known active disease ≥3 years before the first dose of IP and of low potential risk for recurrence

    • Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease

    • Adequately treated carcinoma in situ without evidence of disease
16. Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. hepatitis C, Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA. Testing for HIV is not required at screening but patients with known HIV disease will be excluded from the study.
17. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab or tremelimumab. The following are exceptions to this criterion:

    • Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
    * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
    * Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
18. Receipt of live attenuated vaccine within 30 days prior to the first dose of study drug. NOTE: Patients, if enrolled, should not receive live vaccine whilst receiving study drug and up to 30 days after the last dose of study drug.
19. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab monotherapy or180 days after the last dose of durvalumab + tremelimumab combination therapy.
20. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
21. Prior randomization or treatment in a previous durvalumab and/or tremelimumab clinical study regardless of treatment arm assignment.
22. Has had severe hypersensitivity (≥ Grade 3) to anti -PD1/PDL1 or anti-CTLA4 therapy and/or any of their excipients in the past.
23. Patients who have received prior anti-PD-1, anti-PD-L1 or anti-CTLA-4:

    • Must not have experienced a toxicity that led to permanent discontinuation of prior immunotherapy. All AEs while receiving prior immunotherapy must have completely resolved or resolved to baseline prior to screening for this study.
    * Must not have experienced a ≥Grade 3 immune related AE or an immune related neurologic or ocular AE of any grade while receiving prior immunotherapy. NOTE: Patients with endocrine AE of ≤Grade 2 are permitted to enrol if they are stably maintained on appropriate replacement therapy and are asymptomatic.
    * Must not have required the use of additional immunosuppression other than corticosteroids for the management of an AE, not have experienced recurrence of an AE if re-challenged, and not currently require maintenance doses of > 10 mg prednisone or equivalent per day.
24. Judgment by the investigator that the patient is unsuitable to participate in the study and the patient is unlikely to comply with study procedures, restrictions and requirements.

    -

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2024-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Moh'd Khushman, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
To be determined

RESULTS

PARTICIPANT FLOW:
Groups:
- Novel Combination of Chemotherapy and Immunotherapy: This study has one arm. All enrolled patients will receive a combination of a platinum based chemotherapy regimen (gemcitabine and cisplatin) and a combination of two immune check point inhibitors, anti- CTLA4 (Tremelimumab) and anti PDL-1 (durvalumab).
  Gemcitabine will be administered (gemzar) intravenously, 1000mg/m2 on Day 1 and Day 8 of a 21 day cycle for up to 4 cycles. Cisplatin (Platinol) will be administered intravenously, 25mg//m2 on Day 1 and Day 8 of a 21 day cycle for up to 4 cycles.
  Tremelimumab will be administered intravenously, 300mg flat dose, on Day 1 of cycle 1 only. Durvalumab will be administered intravenously 1500mg on Day 1 of a 21 day cycle for 4 cycles.
  Novel combination of chemotherapy and immunotherapy: This is a study of the combination of platinum based chemotherapy (gemcitabine and cisplatin) and doublet immunotherapy (durvalumab and tremelimumab) in the preoperative setting for intrahepatic cholangiocarcinoma with high risk features. Gemcitabine and cisplatin are chemotherapy agents used in the management of locally advanced and metastatic cholangiocarcinoma. Durvalumab is a programmed cell death ligand 1 (PDL1) blocking antibody, that improves the immune response against cancer. Tremelimumab is an antibody that targets cytotoxic T cell lymphocyte-associated protein 4 (CTLA4) on regulatory T cells. It also improves the immune response against cancer cells
Period: Overall Study
Arm/Group | Novel Combination of Chemotherapy and Immunotherapy
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Novel Combination of Chemotherapy and Immunotherapy
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 43 [43 to 43]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: We will obtain computerized tomography (CT) and/or magnetic resonance imaging (MRI) scans to assess the response to the intervention agents. We are interested in determining the percentage of patients who achieve a complete response or partial response (complete response plus partial response equals to objective response) when treated with intervention agents.
Time Frame: Assessments will occur after 2 cycles (6 weeks) of receiving treatment and after 4 cycles (12 weeks) of receiving treatment or before surgical resection, whichever happens first.
Population: The study terminated prematurely due to slow accrual and study sponsor decision.
Measure: Number; unit: percentage of participants
Arm/Group | Novel Combination of Chemotherapy and Immunotherapy
Number analyzed (Participants) | 1
percentage of participants | 100

2. Secondary Outcome: The Percentage of Participants That Complete Preoperative Therapy
Description: We will assess the percentage of patients who receive all 4 cycles of preoperative therapy
Time Frame: Baseline through 16 weeks of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Novel Combination of Chemotherapy and Immunotherapy
Number analyzed (Participants) | 1
Participants | 1

3. Secondary Outcome: Determine the Safety of the Combination of Intervention Agents by Assessing the Percentage of Patients Who Experience Dose Limiting Toxicities or Develop Adverse Reactions
Description: Adverse reactions will be monitored and documented based on the National Cancer Institute's Common Terminology Criteria for Adverse Events version 5.0. The percentage of patients who experience different grades of adverse events will be assessed
Time Frame: Baseline through 16 weeks of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Novel Combination of Chemotherapy and Immunotherapy
Number analyzed (Participants) | 1
Participants | 1

4. Secondary Outcome: Determine Changes in the Tumor mRNA Gene Expression Pattern, Phenotype of Circulating Cytotoxic T Cells, and Changes in Circulating Markers of Immunogenic Cell Death Following Treatment With Intervention Agents
Description: We will compare the differences in the patterns between the responders and the non responders.
Time Frame: Baseline through 24 months
Population: this was not evaluated on any participants enrolled
Arm/Group | Novel Combination of Chemotherapy and Immunotherapy
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Novel Combination of Chemotherapy and Immunotherapy
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Novel Combination of Chemotherapy and Immunotherapy (N=1)
hospitalization (Gastrointestinal disorders) | 1 (1) — Subject with intrahepatic cholangiocarcinoma was admitted to hospital on 7/3/2023 with Grade 3 vomiting and hypomagnesemia. Started C1D1 on 4/28/23. Last dose drug on 6/9/23. Treated, discharged 7/9/23. Possibly related-Gemcitabine or Cisplatin.

LIMITATIONS AND CAVEATS:
Study sponsor discontinued this study due to low accruals and change in sponsor strategy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-19): https://cdn.clinicaltrials.gov/large-docs/18/NCT04989218/Prot_SAP_000.pdf